CLINICAL TRIAL: NCT03117556
Title: Bilateral Thoracoscopic Splanchnicectomy for Pain Relief in Patients With Unresectable Pancreatic Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no subjects enrolled
Sponsor: University of Louisville (Other)
Collaborators: Norton Healthcare (Other)
Responsible Party: Principal Investigator, Gary C. Vitale, MD, Professor of medicine, General Surgeon, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17.0315
Record Dates: First submitted 2017-04-07; First posted 2017-04-18 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Unresectable Pancreatic Cancer

STUDY DESIGN:
Intervention Model Description: All patients with unresectable pancreatic cancer will be considered for participation in this study. Patients with locally advanced or metastatic cancer that meet inclusion criteria will be randomized into one of two arms, treatment with BTS and narcotic analgesia or treatment with narcotic analgesia alone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BTS Intervention (Experimental): Bilateral thoracoscopic splanchnicectomy and infusaport placement will be performed on patients randomly selected for treatment with BTS and narcotic analgesia. Narcotics will still be prescribed for pain as needed.
  Interventions: Procedure: Bilateral Thoracoscopic Splanchnicectomy
- No BTS Intervention (No Intervention): Patients chosen to be treated with narcotic analgesia alone will undergo infusaport placement only.

INTERVENTIONS:
Procedure: Bilateral Thoracoscopic Splanchnicectomy — BTS will be performed on all patients under general endotracheal anesthesia. Patients will be placed in the prone position. A 5 mm trocar should be placed at the inferior scapular apex on the patient's left side. After confirmation of trocar placement with a 30 degree 5 mm thoracoscope, a second trocar will be placed two intercostal spaces below and two cm medial to the first trocar. After the splanchnic nerves are identified inferior and medial to the sympathetic trunk, the pleura will be incised on both sides of each of the nerves. Skin incisions are then closed and the procedure will then be repeated on the patient's right side.
  Arms: BTS Intervention

SUMMARY:
This study aims to compare the efficacy of bilateral thoracoscopic splanchnicectomy (BTS) to conventional narcotic analgesia for control of abdominal pain in patients with pancreatic ductal adenocarcinoma not amenable to surgical resection.

DETAILED DESCRIPTION:
All patients with unresectable pancreatic cancer will be considered for participation in this study. Patients with locally advanced or metastatic cancer that meet inclusion criteria will be randomized into one of two arms, treatment with BTS and narcotic analgesia or treatment with narcotic analgesia alone. After randomization a baseline pain score will be assessed using the visual analog pain scale. Narcotic dosage and frequency will be evaluated at the time of enrollment. A pre-treatment quality of life score will be recorded using the SF-12® Patient Questionnaire. Patients will also be queried about the presence of nausea and reflux.

After all baseline assessments are complete patients will be taken to the OR to undergo their assigned procedure. BTS and infusaport placement will be performed on patients randomly selected for treatment with BTS and narcotic analgesia. BTS will be performed as described in the study procedure. Patients chosen to be treated with narcotic analgesia alone will undergo infusaport placement only. An evaluation will be completed postoperatively in which the length of stay, post-op complications, and chest X-ray results will be recorded. Follow-up assessments will be conducted 24-48 hours post-procedure and at the time of discharge. Further follow-up assessments will be conducted 14 days, 30 days, and 90 days post-procedure during an office visit with the clinical research team or medical oncology.

ELIGIBILITY:
Inclusion Criteria:

1. Must be 18 years of age
2. Diagnosed with stage III/IV pancreatic cancer
3. Willing and able to comply with the protocol requirements
4. Able to comprehend and have signed the Informed Consent Form (ICF) to participate in the study

Exclusion Criteria:

1. Participating in another clinical trial for the treatment of cancer at the time of screening
2. Pregnant or currently breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2018-04-16 (Estimated); Study Completion 2018-04-16 (Actual)

PRIMARY OUTCOMES:
Abdominal pain | 1 year
  Pain will be measured using a visual analog pain score
Daily Narcotic Requirements | 1 year
  Narcotic usage will be monitored at each follow-up visit

SECONDARY OUTCOMES:
Quality of Life Assessment | 1 year
  Quality of Life will be measured using the SF-12® Patient Questionnaire
Presence of Nausea | 1 year
  Patients will be queried about the presence of nausea using a questionnaire
Presence of Reflux | 1 Year
  Patients will be queried about the presence of reflux using a questionnaire
Use of Anti-emetics | 1 year
  anti-emetic dosage will be measures at each follow-up visit

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Louisville, Louisville, Kentucky
  - Greenville Memorial Hospital, Greenville, South Carolina

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.

REFERENCES:
- [Background] Yadav D, Lowenfels AB. The epidemiology of pancreatitis and pancreatic cancer. Gastroenterology. 2013 Jun;144(6):1252-61. doi: 10.1053/j.gastro.2013.01.068. PMID 23622135
- [Background] Gachago C, Draganov PV. Pain management in chronic pancreatitis. World J Gastroenterol. 2008 May 28;14(20):3137-48. doi: 10.3748/wjg.14.3137. PMID 18506917
- [Background] Katri KM, Ramadan BA, Mohamed FS. Thoracoscopic splanchnicectomy for pain control in irresectable pancreatic cancer. J Laparoendosc Adv Surg Tech A. 2008 Apr;18(2):199-203. doi: 10.1089/lap.2007.0066. PMID 18373443
- [Background] Jones WB, Jordan P, Pudi M. Pain management of pancreatic head adenocarcinomas that are unresectable: celiac plexus neurolysis and splanchnicectomy. J Gastrointest Oncol. 2015 Aug;6(4):445-51. doi: 10.3978/j.issn.2078-6891.2015.052. PMID 26261731
- [Background] Malec-Milewska MB, Tarnowski W, Ciesielski AE, Michalik E, Guc MR, Jastrzebski JA. Prospective evaluation of pain control and quality of life in patients with chronic pancreatitis following bilateral thoracoscopic splanchnicectomy. Surg Endosc. 2013 Oct;27(10):3639-45. doi: 10.1007/s00464-013-2937-0. Epub 2013 Apr 10. PMID 23572221
- [Background] Davis BR, Vitale M, Lecompte M, Vitale D, Vitale GC. An objective study of pain relief in chronic pancreatitis from bilateral thoracoscopic splanchnicectomy. Am Surg. 2008 Jun;74(6):510-4; discussion 514-5. PMID 18556993